CLINICAL TRIAL: NCT07167017
Title: Result Of Karyotyping in Pediatric Patients With Congenital Anomalies and Developmental Delay at Assiut University Children Hospital
Brief Title: Result Of Karyotyping in Pediatric Patients With Congenital Anomalies and Developmental Delay
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manahil Saad Mohamed Elkarsani, Master degree student, Assiut University
Other Study IDs: karyotyping results
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Congenital Anomalies; Development Delay
Keywords: karyotyping; congenital anomalies; developmental delay
MeSH Terms: conditions — Congenital Abnormalities; Learning Disabilities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational cross-sectional study is to study the results of karyotyping analysis for children presented with congenital anomalies and developmental delay aged 1 month to 12 years, the need for further genetic tastings and identification of parents who are carrier of balanced chromosomal translocations. The main question it aims to answer:

What the is the incidence of congenital anomalies tested by karyotyping and the type of chromosomal abnormalities causing the clinical features.

Researcher will take detailed clinical history, physical examination and developmental assessment for children and interpret karyotyping results.

For participants data will be collected regarding:

1. History will be taken including demographic data of child age, parental age, consanguinity and relevant family history and developmental history.
2. Clinical examination for any fascial dysmorphism, congenital heart disease, skeletal deformities, renal anomalies or any associated features.
3. Clinical assessment of developmental milestones.
4. Investigations done including laboratory tests, ultrasound scan, x-rays, CT scan, echocardiography or any other investigation.
5. Karyotyping results detected if aneuploidy or structural abnormality including chromosomal deletions, duplications, translocations or inversions.
6. Other genetics tests done including Comparative microarray, FISH (Fluorescence in Situ Hybridization), and WES (Whole Exome Sequencing).
7. If parental karyotyping for suspected translocations was done.

DETAILED DESCRIPTION:
Chromosomal abnormalities are the leading cause of congenital anomalies with or without neurodevelopmental delay. It is increasing in incidence worldwide and occurs in 10-15% of pregnancies and contributes to 50-70% of spontaneous abortions. The genetic and congenital anomalies are higher in Sub-Saharan Africa by 20% than industrialized countries. Developmental delay (DD) is a measurable lag in achieving the age-related developmental milestones in young children. This could affect one domain (cognitive, motor, speech and language or social) or more than one domain which is global developmental delay. Global Developmental Delay affects 1-3% of children, and the prevalence of intellectual disabilities is estimated to be 18.3/1000 child and adolescent population.

There is limited data of birth prevalence of chromosomal abnormalities in the middle east and Africa. A meta-analysis of 66 articles with 52,569 congenital anomalies cases through Africa showed that the pooled proportion of chromosomal disorders among births with congenital anomalies in Africa is 8.94%, with highest prevalence in North African area than than the other African regions, compared to 12% in the USA. This may indicate underestimation due to limited resources and diagnostic tools in developing countries. This may also contribute to the fact that prevalence in the Middle East and Africa was between 20-30/1000 live births while it was 45-50/1000 live births in developed countries.

Prenatal diagnosis plays an important role in early detection of high-risk infants with congenital anomalies. Cytogenetics tests including karyotyping and Chromosomal Microarray (CMA) are effective prenatal genetic techniques to identify fetal anomalies. This leads to improvement of clinical outcome and performing appropriate genetic counselling. Unbalanced complex chromosomal arrangements (CCRs) is a rare rearrangement that involves three or more chromosomal break points, which mostly is de Novo but can be familial. Carriers of unbalanced CCRs may have Developmental delay and Congenital anomalies while carriers of the balanced type may have recurrent abortions and give birth to children with unbalanced CCRs.

The positive diagnostic yield of G-banded karyotyping with its inability to detect chromosomal abnormalities less than 10 Mb was 7.4% after exclusion of Down Syndrome detection, compared CMA in detecting chromosomal abnormalities in patients with unexplained developmental delay, Autistic spectrum disorders and multiple congenital anomalies which is 15-20%. This due to the high resolution of CMA and ability to detect smaller chromosomal aberrations. There was a high association between presence of hypotonia and diagnostic karyotyping (p.value=<0.001) (8), so despite the superiority of CMA in detecting small deletions and duplications it is recommended to reserve karyotyping for patients with obvious chromosomal syndromes (e.g., Down syndrome), a family history of chromosomal rearrangement, or a history of multiple miscarriages.

Another evidence which leads to recommendation to make CMA is first tier test for with developmental delay, intellectual disability, autism spectrum disorder, and/or multiple congenital anomalies, that the prevalence of congenital anomalies caused by microdeletions and duplications is about 1.2% compared to 0.2% caused by trisomies (21,13,18). CMA is cost-effective in diagnosing Developmental delay and Congenital anomalies than karyotyping as well as when testing the parents in case of copy number variant of unknown significance, but its use is limited by its higher cost. Karyotyping remains a test with a reasonable diagnostic yield for countries with limited resources. Further genetic tests may be required to diagnose patients where karyotyping and CMA fails to detect a chromosomal abnormality or a pathologic copy number of variants. This includes whole exome sequencing (WES) and targeted gene panels for intellectual disabilities which includes 1,252 genes. Leite A, et al. found a diagnostic rate of 42,3% when using the three diagnostic methods of karyotyping, CMA and WES.

G-banded Karyotyping and molecular karyotyping (CMA) may impact the clinical outcome of the patient in many aspects, this includes reaching a diagnosis, predicting outcome and level of care and multidisciplinary team assigned for managing the affected patients. It is mandatory to establish an effective cytogenetic-diagnostic facility beside well-trained genetic counsellors. This is in addition to developing a local registry system for congenital anomalies. On the other hand, parents testing and prenatal counselling or antenatal genetic testing in cases of balanced chromosomal rearrangements carriers is mandatory towards preventing recurrence.

ELIGIBILITY:
Inclusion Criteria:

All patients aged between 1 month to 12 years old who are presented with morphologic congenital anomalies associated with developmental delay either global DD or isolated developmental domain (cognitive, motor, speech and language or social) who are tested for chromosomal abnormalities

Exclusion Criteria:

Any patient aged between 1 month and 12 years old who is presented with Developmental Delay and congenital anomalies who didn't undergo karyotyping or other genetic testing.

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged between 1 months, and 12 years presented at Assiut university hospital with congenital anomalies and developmental delay either global developmental delay or affecting one domain (cognitive, motor, speech and language or social) during the year 2025-2026.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Result Of Karyotyping in Pediatric Patients with Congenital Anomalies and Developmental Delay at Assiut University Children Hospital | November 2025-December 2026
  To detect the incidence of congenital anomalies and developmental delay tested with karyotyping and to detect karyotyping findings of chromosomal numerical or structural abnormalities that cause clinical features.

SECONDARY OUTCOMES:
Result Of Karyotyping in Pediatric Patients with Congenital Anomalies and Developmental Delay at Assiut University Children Hospital | November 2025-December 2026
  To determine patients requiring further testing due to inability of karyotyping in reaching a diagnosis
  - Detect parents requiring karyotyping to detect carriers of balanced chromosomal translocations

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mahrous Mohamed, Professor of pediatrics, Study Director — Assiut University; Mohamed Abobakr Mohamed, Lecturer of pediatr, Study Director — Assiut University